CLINICAL TRIAL: NCT05105295
Title: Immunogenicity and Safety of a Third Dose and Immune Persistence of BBIBP-Corv Vaccine in People With Human Immunodeficiency Virus Infected
Brief Title: Immunogenicity and Safety of a Third Dose and Immune Persistence of BBIBP-Corv Vaccine in People With HIV Infected
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BIBP2021HIV-third dose
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; HIV Infections
MeSH Terms: conditions — COVID-19; HIV Infections

STUDY DESIGN:
Intervention Model Description: Subjects aged ≥18 with infected with HIV who have completed the schedule of two doses for 3 months receive a third dose of inactivated COVID-19 vaccine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Subjects receive a third dose of inactivated COVID-19 vaccine
  Interventions: Biological: Inactivated COVID-19 vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 vaccine — receive a third dose of inactivated COVID-19 vaccine

SUMMARY:
Evaluation of immunogenicity, safety and persistence of the subjects with HIV infected received the third dose of inactivated COVID-19 vaccine .

DETAILED DESCRIPTION:
The subjects aged ≥18 years with HIV infected who have completed the schedule of two doses for 3 months recruited to receive a third dose of inactivated COVID-19 vaccine.

Blood samples will be collected 3 times: before the third dose of vaccinatioin，28 days and 6 months after the third dose of vaccination.

Any local or systemic adverse events that occurred within 21 days after vaccination will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18.
* Body temperature < 37.3 ° C confirmed by clinical examination before enrollment .
* Subjects who meet the diagnostic criteria for HIV infection and AIDS.
* CD4+ count is less than 500/ul and more than 50/ul .
* Female subjects of reproductive age declare that they are not pregnant, have no birth plan in the first 3 months after enrollment, and have taken effective contraceptive measures in the first 2 weeks before enrollment.
* Able and willing to complete the entire study plan during the study follow-up period.
* Have the ability to understand the study procedures, voluntarily sign informed consent, and comply with the requirements of the clinical study protocol.
* Subjects participating in the past clinical trial have completed two doses of COVID-19 vaccine and blood collection before and after immunization;

Exclusion Criteria:

* Subjects were previously confirmed cases of COVID-19 or asymptomatic infected persons.
* Being allergic to any component of vaccines (including excipients) .
* Subjects who have experienced severe allergic reactions to vaccines (e.g. acute anaphylaxis, urticaria, angoneeurotic edema, dyspnea, etc.).
* Having uncontrolled epilepsy and other progressive neurological disorders and a history of Guillain-Barre syndrome.
* Injection of non-specific immunoglobulin within 1 month before enrollment.
* Pregnant and lactating women.
* The subjects are suffering from an acute illness; Or thrombocytopenia patients with platelet count < 20×10^9/L within three days before inoculation, that is, patients at high risk of spontaneous bleeding.
* Acute HIV infection and opportunistic infection.
* Subjects with co-opportunistic infections who did not receive antiviral therapy.
* Subjects with CD4+ count less than 50/ul who have not received antiviral therapy.
* HIV-infected subjects undergoing treatment with severe drug interactions and overlapping toxicity (kidney damage, liver damage, hematological problems, etc.).
* Patients with malignant tumors are undergoing chemotherapy and radiotherapy before and after surgery.
* Subjects who had vaccine-related adverse reactions after the second dose.
* Having high fever (axillary temperature ≥39.0℃) for three days after the second dose of inoculation, or severe allergic reaction.
* Having any adverse nervous system reaction after the second dose.
* Other subjects whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 28 days after the 3th dose (Day 28)
  The rate of seroconversion against coronavirus
Neutralizing antibody level | Before the 3th dose (Day 0)
  Neutralizing antibody GMT against coronavirus before the 3th dose
Neutralizing antibody level | 28 days after the 3th dose (Day 28)
  Neutralizing antibody GMT against coronavirus after the 3th dose
Neutralizing antibody level | 6 months after the 3th dose
  Neutralizing antibody GMT against coronavirus after the 3th dose

SECONDARY OUTCOMES:
Adverse events rate | 0-21days following vaccinations
  Analyse the incidence of adverse events following vaccination, both solicited and unsolicited
Serious adverse event rate | 0-6 months
  Report and analyse serious adverse events
T cell count | before the 3th dose (Day 0)
  T cell count （CD4+T，CD8+T，etc.）
T cell count | 28 days after the 3th dose (Day 28)
  T cell count （CD4+T，CD8+T，etc.）
HIV viral load | before the 3th dose (Day 0)
  HIV viral load
HIV viral load | 28 days after the 3th dose (Day 28)
  HIV viral load

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang provincial center for disease control and prevention, Hangzhou, Zhejiang, China